CLINICAL TRIAL: NCT06265207
Title: The Effect of Virtual Reality Applied to Women Before Mammography on Pain, Anxiety and Satisfaction Level: Single-Blind Randomized Controlled Study
Brief Title: The Effect of Virtual Reality on Pain, Anxiety and Satisfaction Level Before Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Collaborators: Kafkas University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ArdahanU-Simsekli-DS-02
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-02

CONDITIONS: Mammography; Early Diagnosis of Cancer
Keywords: Mammography; virtual reality; pain; anxiety; satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Single Blind Parallel Group Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the researcher will be conducting the research, blinding will not be possible, and separate consent forms were prepared for the experimental and control groups, without specifying which group they were in, and it was planned to blind the participants in this way. In addition, in order to prevent statistical bias, it is planned to prevent bias in data analysis by coding the data as first group and second group, rather than experimental and control group, when entering the data into SPSS, and by not giving information about which group is the experiment and which is the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Before the mammography, a 20-minute relaxing video featuring nature and forest views will be watched with VR SHINECON 360 degree glasses. Since it is seen in the literature that watching a video for 20 minutes provides effective results, the video viewing time was determined as 20 minutes.
  Interventions: Other: Virtual reality
- Control group (Active Comparator): No additional application to routine procedures will be applied to the control group.
  Interventions: Other: routine maintenance

INTERVENTIONS:
Other: Virtual reality — Before the mammography, a 20-minute relaxing video featuring nature and forest views will be watched with VR SHINECON 360 degree glasses. Since it is seen in the literature that watching a video for 20 minutes provides effective results, the video viewing time was determined as 20 minutes.
  Arms: Experimental group
Other: routine maintenance — routine maintenance
  Arms: Control group

SUMMARY:
In this study, it is planned to determine the effect of virtual reality applied to women before mammography on pain, anxiety and satisfaction levels. For this purpose, individuals applying for breast cancer screening will first be randomly divided into experimental and control groups. Pain, anxiety and satisfaction level evaluation forms will be applied to the experimental group before the mammography procedure. A relaxing video will be watched with virtual reality glasses and the mammography will be performed. At the end of the mammography, the relevant forms will be applied to the individuals again. The control group will not be subjected to any additional application that will continue with the applied routine.

DETAILED DESCRIPTION:
Purpose and duration of the research: This research is to determine the effect of virtual reality applied to women before mammography on the pain, anxiety and satisfaction levels.

Materials and methods of the research: This research is planned to be carried out in a pre-test post-test single-blind randomized controlled experimental design.

Research Questions/Hypotheses:

Hypotheses of the Research H0: Virtual reality applied to women before mammography has no effect on pain, anxiety and satisfaction levels.

H1a: Virtual reality applied to women before mammography has an effect on pain. H1b: Virtual reality applied to women before mammography has an effect on anxiety.

H1c: Virtual reality applied to women before mammography has an effect on the satisfaction level.

Dependent variables of the research; these are the scores to be taken from the Visual Comparison Scale, State Anxiety Inventory and Satisfaction Rating Scale. The independent variable of the research is; This is a video that will be watched with virtual reality glasses.

The research was planned to be carried out in the Cancer Early Diagnosis, Screening and Education Center (Ketem) unit. Individuals who applied to Kars Provincial Health Directorate KETEM Unit during the research process will constitute the population of the research. A power analysis was performed to determine the sample size of the study, and accordingly, with a Cohen-d effect size of 0.80 (Goulet-Pelletier & Cousineau, 2018; Kilic, 2014), a power of 0.95, an alpha margin of error of 0.05, the minimum sample size planned to be included in the study was 35 for the experimental group, It was determined that there should be a total of 70 participants, 35 in the control group. Considering the 10% loss, it is planned to include four more patients in each group, making a total of 78 participants the sample of the study.

Randomization and blinding The block randomization method was chosen in the study to eliminate selection bias and distribute participants equally to the groups. After determining the participants who meet the inclusion and exclusion criteria, a pre-test was applied to those who voluntarily agreed to participate, and then they will be randomized into experimental and control groups. 78 participants who met the research criteria were assigned to groups by block randomization. It will be decided which group is the experiment and which group is the control, by a lottery drawn by a nurse independent of the study before the implementation.

Descriptive Information Form, Visual Comparison Scale, State Anxiety Inventory and Satisfaction Evaluation Scale will be used as data collection tools.Visual Comparison Scale; It provides a simple assessment of pain. Pain is rated between mild pain = 0 and unbearable pain = 10. Pain intensity is categorized as 1-3 mild, 4-6 moderate, and 7-10 severe.

State Anxiety Inventory; It was developed by Spielberger et al. to evaluate the anxiety level of individuals. The scale measures trait and state anxiety. In this study, 20 items that evaluate state anxiety will be used to evaluate state anxiety. The scale is scored in a four-point Likert type, as "1 = not at all, 2 = a little, 3 = a lot and 4 = completely". The score obtained shows the state anxiety score. The lowest score that can be obtained from the scale is 20, while the highest score is 80. A high score indicates high anxiety, while a low score indicates low anxiety level.

Satisfaction Evaluation Scale; It is a scale that individuals can easily understand and is easy to apply. It is a scale indicated by a horizontal or vertical line, ranging from 0 = not at all satisfied to 10 = quite satisfied. The evaluation is made based on the average value.

ELIGIBILITY:
Inclusion Criteria:

* Having applied for mammography for screening purposes,
* having no communication problems,
* being over 18 years of age,
* not having a history of breast cancer
* voluntarily agreeing to participate in the study

Exclusion Criteria:

* Being screened for breast cancer
* having vision or hearing problems
* being under 18 years of age.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female applicants will be included due to breast cancer screening.
Enrollment: 78 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Visual Comparison Scale | an average of 6 months after the completion of the initiative
  It provides a simple assessment of pain. Pain is rated between mild pain = 0 and unbearable pain = 10. Pain intensity is categorized as 1-3 mild, 4-6 moderate and 7-10 severe.
State Anxiety Inventory | an average of 6 months after the completion of the initiative
  The scale measures trait and state anxiety. In this study, 20 items that evaluate state anxiety will be used to evaluate state anxiety. The scale is scored in a four-point Likert type, as "1 = not at all, 2 = a little, 3 = a lot and 4 = completely". The lowest score that can be obtained from the scale is 20, while the highest score is 80. A high score indicates high anxiety, while a low score indicates low anxiety level.
Satisfaction Evaluation Scale | an average of 6 months after the completion of the initiative
  It is a scale that individuals can easily understand and is easy to apply. It is a scale indicated by a horizontal or vertical line, ranging from 0 = not at all satisfied to 10 = quite satisfied. The evaluation is made based on the average value.

CONTACTS AND LOCATIONS:
Overall Officials: Derya ŞİMŞEKLİ, Lecturer, Principal Investigator — Ardahan University
Locations (1):
- Cancer Early Diagnosis, Screening and Education Center Unit, Kars, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No